## IZMIR KÂTIP ÇELEBI UNIVERSITY SOCIAL RESEARCH ETHICS COMMITTEE INFORMED VOLUNTEER CONSENT FORM

It will be held by Fatih Esad Topal and Emine Oruç. We invite you to the research titled "The value of endtidal capnography in the evaluation of mortality and morbidity in patients who apply to the emergency department with complaints of gastrointestinal bleeding." The scope and purpose of this study is to measure the carbon dioxide pressure in the breath of a patient who applied to the emergency department due to gastrointestinal bleeding by breathing with a special mask. It will be investigated whether this measured value is associated with gastrointestinal bleeding and whether it affects the course of the disease. The measurement of end tidal carbon dioxide value with a capnometer is done by breathing normally with a mask attached to you (your patient). Your (patient's) treatment will not be disrupted in any way. No invasive procedure will be performed on you (your patient) for this measurement. Approximately 2 minutes will be required for this study. You are asked to separate. Participating in this study is entirely voluntary. You will not be asked for any fee to participate in this study, and you will not be paid for participating. In order to achieve the purpose of the study, you are expected to answer all the questions completely, sincerely, in the way that best suits you, without being under anyone's pressure or suggestion. Reading/having it read to you and approving this form means that you agree to participate in the research. However, you also have the right not to participate in the study or to withdraw at any time after agreeing to participate. The information obtained from this study will be used entirely for the purpose of the research and your personal information will be kept confidential. If you need more information other than this information about the purpose of the research, you can ask the researcher now or request information by e-mail at dreminekilincc@gmail.com or by phone at 05386162340.

Thank you for your interest in the research.

Researcher's

Name-Surname: Emine Oruc

Signature:

History:01.06.2020

Contact Information: E-mail:dreminekilincc@gmail.com

Phone:05386162340

## PARTICIPANT STATEMENT

I have read / ensured that the information above, which should be given to the participant before the research, was read. Written and verbal explanations about the study were made by the researcher/researchers named below. I understood the scope and purpose of the study in which I was asked to participate and my responsibilities as a volunteer. I was explained the possible risks and benefits of the study. Adequate assurance was given that my personal information would be carefully protected.

Under these conditions, I agree to participate in this research voluntarily, without any pressure or suggestion.

I was given a signed copy of this form.

Participant:
Name-Surname:
Signature:

History:

Contact Information: E-mail:

Phone: